CLINICAL TRIAL: NCT03803358
Title: The Effects of Non-invasive Ventilation During Cycle Exercise Within a 3-week Pulmonary Rehabilitation Program in COPD Patients With Chronic Hypercapnic Respiratory Failure - a Randomized Controlled Trial
Brief Title: NIV-Training in Hypercapnic COPD Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Schön Klinik Berchtesgadener Land (Other)
Collaborators: Löwenstein Medical GmbH & Co. KG (Unknown); Bad Reichenhaller Forschungsanstalt (Unknown)
Responsible Party: Principal Investigator, Klaus Kenn, Prof. Dr. Klaus Kenn, Schön Klinik Berchtesgadener Land
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NIV-Training
Record Dates: First submitted 2019-01-07; First posted 2019-01-14 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: COPD
Keywords: CHRF; NIV; exercise training
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Exercise; Noninvasive Ventilation

STUDY DESIGN:
Intervention Model Description: A total of 26 COPD patients in GOLD Stages IV diagnosed with CHRF, already treated with nocturnal NIV and referred for a comprehensive PR program will be recruited and randomized into two groups: 1) exercise with NIV during exercise (nocturnal NIV will continue) and 2) control group - exercise without NIV during exercise (nocturnal NIV will continue).
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cycle exercise with additional NIV (Experimental): In the intervention group (exercise training with non-invasive ventilation) exercise NIV pressures will be optimally adjusted to each individual patient to decrease TcPCO2 values. An IPAP of at least 15 cmH20 will be used to provide sufficient pressure to relief patients breathing muscles. Nocturnal NIV will be continued.
  Interventions: Other: exercise training with non-invasive ventilation
- cycle exercise without NIV (Active Comparator): In the control Group (standard exercise training without NIV ), patients will be execute cycle exercise without additional NIV (usual care). Nocturnal NIV will be continued.
  Interventions: Other: standard exercise training without NIV

INTERVENTIONS:
Other: exercise training with non-invasive ventilation — In the intervention group (exercise training with non-invasive ventilation) exercise NIV pressures will be optimally adjusted to each individual patient to decrease TcPCO2 values. An IPAP of at least 15 cmH20 will be used to provide sufficient pressure to relief patients breathing muscles. Nocturnal NIV will be continued.
  Arms: cycle exercise with additional NIV
Other: standard exercise training without NIV — In the control Group (standard exercise training without NIV ), patients will be execute cycle exercise without additional NIV (usual care). Nocturnal NIV will be continued.
  Arms: cycle exercise without NIV

SUMMARY:
The aim of the study is to investigate the additional effects of the use of NIV during exercise within a 3-week PR program on exercise capacity in COPD patients with chronic hypercapnic respiratory failure.

DETAILED DESCRIPTION:
Scientific Background/ Rationale:

Quality of life and exercise tolerance are commonly reduced in people with chronic obstructive pulmonary disease (COPD), especially in people with chronic hypercapnic respiratory failure (CHRF). Endurance exercise training as part of a pulmonary rehabilitation (PR) programme is an important treatment for people with COPD and has been shown to improve quality of life, exercise tolerance and physical activity. However, individuals with CHRF may have difficulties performing endurance exercise at an adequate training intensity to achieve the desired physiological changes.

Non-invasive ventilation (NIV) is a method of providing breathing support using a ventilator and is usually delivered via a full face mask. A recent study showed that during a single exercise session in people with CHRF, NIV dramatically improves exercise tolerance and reduces breathlessness. Consequently, NIV used over a complete exercise training program may allow people with COPD and CHRF to exercise at a higher intensity to achieve greater improvement in exercise tolerance, quality of life and physical activity. So far this has only been tested in a small number of studies with small numbers of participants, and none with CHRF. It is currently not known from literature whether the demonstrated benefits of NIV during exercise training are clinically worthwhile or cost-effective.

Aims The aim of the study is to investigate the additional effects of the use of NIV during exercise within a 3-week PR program on exercise capacity in COPD patients with chronic hypercapnic respiratory failure.

Hypothesis It is assumed that a 3-week exercise training program with additional NIV, using titrated pressures, reduces the work of breathing. With this, it is theorized, COPD patients with CHRF are able to train for a longer duration and/ or with higher training intensities over the course of the training program and may achieve better PR outcomes.

Primary Hypothesis:

H.0: COPD-Patients with CHRF have the same increase in exercise capacity (endurance cycle time) when training with additional NIV as without NIV, during a 3-week PR program.

H.1: COPD-Patients with CHRF have a superior increase in exercise capacity (endurance cycle time) when training with additional NIV as without NIV, during a 3-week PR program.

Main Objective To determine if NIV during exercise is a useful tool for increasing exercise tolerance in hypercapnic patients, exercise tolerance (cycle endurance time) will be measured without NIV at PR admission/ discharge

Materials and Method A total of 26 COPD patient (age: 40-80 years) in GOLD Stages IV diagnosed with CHRF, already treated with nocturnal NIV and referred for a comprehensive PR program will be recruited and randomized into two groups: 1) exercise with NIV during exercise (nocturnal NIV will continue) and 2) control group - exercise without NIV during exercise (nocturnal NIV will continue).

Initially, patients will perform a maximum cardiopulmonary test to determine the Peak Work Rate (WRpeak). On a separate day, patients will perform a cycle endurance test (CET) at 75%WRpeak without NIV using oxygen as prescribed, if needed. TcPCO2, heart rate and SpO2 via SenTec will be measured continuously during CET. In addition to the continuously recorded data, dyspnoea/ respiratory effort/ leg-fatigue (10-point Borg scale), capillary blood gases and the arterial blood pressure will be taken at the beginning/ end/ recovery/ isotime of the CET.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of very severe COPD Gold Stage IV
* Age: 40-80 years
* PaCO2 >50mmHg (at rest, during sleep or exercise)
* Implemented nocturnal non-invasive ventilation therapy

Exclusion Criteria:

* Concomitant cardiovascular, orthopaedic or neurological conditions that are likely to be the primary impairment to exercise performance
* Other significant pulmonary disease which could affect exercise or NIV (e.g. asthma)
* BMI > 35 kg/m2
* Inability to give informed consent

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-01-07 (Actual); Primary Completion 2021-07-27 (Actual); Study Completion 2021-07-27 (Actual)

PRIMARY OUTCOMES:
Exercise tolerance | Day 1 and Day 21
  Change in cycle endurance time without NIV within PR

SECONDARY OUTCOMES:
Partial pressure of transcutaneous carbon dioxide | Day 1 and Day 21
  Change in partial pressure of carbon dioxide levels during CET, recorded via SenTec (Switzerland, Therwill)
Oxygen saturation | Day 1 and Day 21
  Change in Oxygen Saturation during CET, recorded via SenTec (Switzerland, Therwill)
Heart rate | Day 1 and Day 21
  Change in Heart Rate during CET, recorded via SenTec (Switzerland, Therwill)
Partial pressure of carbon dioxide | Day 1 and Day 21
  Change in partial pressure of carbon dioxide pre/ post CET, recovery, isotime, recorded via capillary taken blood gases
Partial pressure of oxygen | Day 1 and Day 21
  Change in partial pressure of oxygen pre/ post CET, recovery, isotime, recorded via capillary taken blood gases
Arterial blood pressure | Day 1 and Day 21
  Change in arterial blood pressure pre/ post CET, recovery, isotime
Patients perception - Dyspnoe | Day 1 and Day 21
  Change in perceived dyspnoea /respiratory effort pre/ post CET, recovery, isotime recorded via Borg Scale
Patients perception - leg fatigue | Day 1 and Day 21
  Change in perceived leg fatigue pre/ post CET, recovery, isotime recorded via Borg Scale
Patients Quality of life - Chronic Respiratory Questionnaire | Day 1 and Day 21
  Change in Chronic Respiratory Questionnaire
Patients Quality of life - Severe Respiratory Insufficiency Questionnaire | Day 1 and Day 21
  Change in Severe Respiratory Insufficiency Questionnaire
Anxiety and Depression | Day 1 and Day 21
  Change in Hospital Anxiety and Depression Scale
Maximal voluntary muscle contraction | Day 1 and Day 21
  Change in muscle contraction force (m. rectus femoris) recorded via MicroFet
Patients perception to physical Training with additional NIV | Day 1 and Day 21
  Patients in the Intervention Group will be interviewed how they perceived the Treatment, via a questionnaire with open- and closed ended questions

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Kenn, Prof. Dr., Principal Investigator — Philipps University of Marburg, Department of pulmonary rehabilitation
Locations (1):
- Schoen Klinik Berchtesgadener Land, Schönau am Königssee, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schneeberger T, Dennis CJ, Jarosch I, Leitl D, Stegemann A, Gloeckl R, Hitzl W, Leidinger M, Schoenheit-Kenn U, Criee CP, Koczulla AR, Kenn K. High-intensity non-invasive ventilation during exercise-training versus without in people with very severe COPD and chronic hypercapnic respiratory failure: a randomised controlled trial. BMJ Open Respir Res. 2023 Nov 22;10(1):e001913. doi: 10.1136/bmjresp-2023-001913. PMID 37993279